CLINICAL TRIAL: NCT00614549
Title: Long-term Evaluation of the Efficacy and Safety of Levetiracetam in Routine Clinical Practice in the Czech and Slovak Republics, Hungary, and Romania - Non-interventional Study
Brief Title: Efficacy and Safety of Levetiracetam in Routine Clinical Practice in Czech and Slovak Republics, Hungary, and Romania.
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: N01283
Record Dates: First submitted 2008-01-11; First posted 2008-02-13 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Epilepsy
Keywords: Levetiracetam; Keppra; Epilepsy; Efficacy; Safety
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Levetiracetam: Patients treated with Levetiracetam

SUMMARY:
To evaluate, over 1 year period, the efficacy and safety of newly prescribed levetiracetam as add-on treatment (POS, myoclonoc seizures in JME and PGTCS in IGE) or primary monotherapy (partial onset seizures) in adult and paediatric patients within the approved age limits in routine clinical practice in Czech and Slovak Republics, Hungary, and Romania. Non-interventional study.

ELIGIBILITY:
Inclusion Criteria:

* diagnoses of partial onset seizures (POS) with or without secondary generalisation or Juvenile Myoclonic Epilepsy (JME) or another IGE with PGTCS
* newly prescribed levetiracetam as add-on treatment (POS, myoclonic seizures in JME and PGTCS in IGE) or monotherapy (partial onset seizures only) in newly diagnosed patients. Newly prescribed means inclusion of the patients in whom a decision has been made to prescribe LEV and the first dose is just to be prescribed.
* age 4 years or above for partial onset seizures, 12 years or above for MS in JME or PGTCS in IGE, 16 years or above for monotherapy
* patient written informed consent

Exclusion Criteria:

* indications other than those defined in inclusion criteria
* history of allergic or anaphylactic reactions to levetiracetam or other pyrrolidone derivatives and excipients included

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinics and hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 2569 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Retention rate after 6 and 12 months | 6 and 12 months

SECONDARY OUTCOMES:
Seizure freedom for the last 6 and 12 months | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)